CLINICAL TRIAL: NCT06655285
Title: The Impact of Tumor-associated Inflammatory Adhesion on the Prognosis of Colon Cancer Patients: a Study Based on the SEER and Chinese Multi-center Databases
Brief Title: The Impact of Inflammatory Adhesion on the Prognosis of Colon Cancer Patients
Status: Completed | Type: Observational
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Jianqiang Tang, Associate professor, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Other Study IDs: NCC3650
Record Dates: First submitted 2024-10-22; First posted 2024-10-23 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-11

CONDITIONS: Colon Cancer
Keywords: Colon Cancer; Prognosis; Tumor-associated inflammatory adhesion
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- the U.S. National Cancer Center SEER database: SEER*Stat software (version 8.4.3) collected 17 registries cohort data on colon cancer patients between 2010 and 2019.
  Interventions: Other: This was a retrospective study and no patient intervention was performed.
- Chinese multi-center database: Chinese multi-center database includes patients from January 2010 to December 2021 at 3 institutions.
  Interventions: Other: This was a retrospective study and no patient intervention was performed.

INTERVENTIONS:
Other: This was a retrospective study and no patient intervention was performed. — This was a retrospective study and no patient intervention was performed.

SUMMARY:
The purpose of this study is to explore the impact of tumor-associated inflammatory adhesion on the prognosis of colon cancer patients.

DETAILED DESCRIPTION:
In some colon cancer patients, although adhesions between the tumor tissue and surrounding organs are found during surgery, postoperative pathology confirms that the tumor has not directly invaded the adhered organs; instead, the adhesions are caused by tumor-associated inflammation. This condition is defined as tumor-associated inflammatory adhesion.

Currently, the impact of tumor-associated inflammatory adhesion on patient prognosis is still unclear. This study aims to explore the impact of tumor-associated inflammatory adhesion on the prognosis of colon cancer patients through the Surveillance, Epidemiology, and End Results (SEER) and Chinese multi-center databases.

ELIGIBILITY:
Inclusion Criteria:

1. The patient was pathologically diagnosed as colon adenocarcinoma by endoscopic biopsy before operation.
2. All patients were considered to have tumors invading adjacent organs during surgery
3. All patients underwent radical surgery.

Exclusion Criteria:

1. Patients with distant metastasis, recurrent colon cancer and pT4b CRC were excluded.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study utilized the Chinese multi-center database as well as the SEER 17 registries database. The Chinese multi-center database contains data of patients between January 2010 and December 2021, at 3 institutions. SEER*Stat software (version 8.4.1.1) was used for collecting 17 registries cohort data on patients diagnosed with NMIBC between 2010 and 2019.
Sampling Method: Non-Probability Sample
Enrollment: 229 (Actual)
Dates: Start 2024-10-24 (Actual); Primary Completion 2024-10-26 (Actual); Study Completion 2024-10-27 (Actual)

PRIMARY OUTCOMES:
Overall survival time (OS) | up to 10 years
  OS, defined as the time from the first diagnosis to death from any cause or the last follow-up for surviving patients
Cancer-specific survival time (CSS) | up to 10 years
  CSS refers to the duration from diagnosis of a tumor until the patient succumbs to the tumor, excluding deaths from other causes.
Recurrence free survival time (RFS) | up to 10 years
  RFS is the time from the time a patient achieved R0 resection after surgery to the time of recurrence or the end of follow-up.

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China